CLINICAL TRIAL: NCT01470261
Title: Attention Deficit Hyperactivity Disorder Drugs Use Chronic Effects
Acronym: ADDUCE
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Collaborators: Zentralinstitut für Seelische Gesundheit Mannheim (Other); Universita degli Studi di Cagliari (Unknown); Vadaskert Child and Adolescent Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Sarah Inglis, Trial Manager, University of Dundee
Other Study IDs: 2011PW02
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: methylphenidate; ritalin; Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ADHD medicated: Children aged 5-17 years with clinical diagnosis of ADHD and not previously treated with methylphenidate who have an agreement with their physician to begin treatment with methylphenidate.
- ADHD unmedicated controls: Children aged between 5-17 years with clinical diagnosis and not previously treated with methylphenidate who have an agreement with their physician NOT to treat with methylphenidate
- Non-ADHD controls: Any child, including siblings of a child in either the ADHD-medicated or ADHD-unmedicated control group, who is 5-17 years old. These children must have a low rating (<1.5) on the clinician-rated Swanson Nolan and Pelham IV Rating scale (SNAP IV) and not be medicated with with either dexamfetamine or atomoxetine.

SUMMARY:
The aim of the ADDUCE project is to investigate any adverse effects of methylphenidate (trade name ritalin) on growth, neurological system, psychiatric states and cardiovascular system over a two year period in children and adults.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders in children, affecting approximately 5% children in Europe. Methylphenidate (MPH, trade name ritalin) is the most-commonly prescribed medication for ADHD children; it is also increasingly used in ADHD adults. In 2007, the European Commission requested a referral to the Committee for Medicinal Products for Human Use (CHMP) under Article 31 of Directive 2001/83/EC, as amended, for MPH because of safety concerns. The CHMP concluded that study of the long-term effects of MPH on growth, sexual development, neurological system, psychiatric states and cardiovascular system is needed. In response to the CHMP s concerns, the ADDUCE (Attention Deficit Hyperactivity Disorder Drugs Use Chronic Effects) research team has been formed by a consortium of experts in the fields of ADHD, drug safety, neuro-psychopharmacology and cardiovascular research.

The ADDUCE project aims to investigate the long-term adverse effects of MPH on growth, neurological system, psychiatric states and cardiovascular system in children and adults.

Furthermore the ADDUCE team will develop research tools for the evaluation of adverse effects of MPH on cognition and motivation.

ELIGIBILITY:
Inclusion Criteria:

ADHD-treated group:

* Clinical diagnosis of ADHD
* Aged between 5 and 17 years.
* Not previously treated with methylphenidate
* Agreement between clinician, patient and their family to commence on methylphenidate (baseline measures will be taken before first prescription of methylphenidate is issued).
* Any co-medication other than dexamfetamine or atomoxetine will be allowed.
* All psychiatric and physical illness comorbidities will be allowed

ADHD-unmedicated controls:

* Clinical diagnosis of ADHD not previously treated with medication.
* Aged between 5 and 17 years.
* Agreement between clinician, patient and their family not to treat with methylphenidate.
* Any medication other than dexamfetamine or atomoxetine will be allowed.
* All comorbidities will be allowed.

Non-ADHD controls:

* Child who does not have ADHD.
* Aged between 5 and 17 years.
* Mean total clinician rated Swanson Nolan and Pelham IV Rating scale (SNAP IV) score (ADHD items) < 1.5
* Parent rated Strengths and Difficulties Questionnaire (SDQ) Hyperactivity Score within normal range for country (e.g. < 6 for UK)
* Any current medication other than dexamfetamine or atomoxetine will be allowed.
* Must never have taken methylphenidate
* Any other mental health or physical illness diagnoses will be allowed.

Exclusion Criteria:

All Groups:

* Current or past treatment with dexamfetamine or atomoxetine.

Un-medicated ADHD controls:

* Previous or current treatment with methylphenidate.

Non-ADHD controls:

* Previous or current treatment with methylphenidate.
* Clinician rated SNAP score ≥ 1.5. Parent rated SDQ Hyperactivity Score in Borderline or Abnormal range.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Attention Deficit Disorder clinic
Sampling Method: Probability Sample
Enrollment: 1398 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The height velocity standard deviation score | 2 years
  Child's height velocity-mean height velocity for sex and age / Standard deviation of height velocity for sex and age.

SECONDARY OUTCOMES:
Changes in growth | 2 years
  * Proportion height < 2nd centile, 0.4th centile (according to best available country specific norms)
  * Weight (z-scores according to best available country specific norms)
  * Proportion weight < 2nd centile, 0.4th centile (according to best available country specific norms)
  * BMI (z-scores according to best available country specific norms)
  * Proportion BMI < 2nd centile, 0.4th centile (according to best available country specific norms)
  * Pubertal stage (Tanner stage)
  * Bone age (selected sample from Italian cohort)
Changes to the cardiovascular system | 2 years
  * Heart rate
  * Proportion heart rate > 120 bpm
  * Diastolic blood pressure
  * Proportion diastolic blood pressure > 90 mm/hg
  * Systolic blood pressure
  * Proportion systolic blood pressure > 95th centile
Effects on Psychiatric state | 2 years
  * SNAP-IV mean scores
  * Clinical Global Impressions score(CGI; severity, improvement)
  * Children's Global Assessment Scale score (CGAS)
  * Strengths and Difficulties questionnaire (SDQ)
  * Mood and Feelings Scale (parent and child ratings)
  * Developmental and Wellbeing Assessment
  * DAWBA Rapidly changing mood section (proportion > cut off)
  * DAWBA tics section (proportion > cut off)
  * Columbia - Suicide Severity Rating Scale
  * Psychosis-like symptoms
  * Substance Use Questionnaire
Changes in neurological state | 2 years
  * Child's Sleep Habits Questionnaire (CSHQ; total score and subscale scores, proportion > cut offs)
  * Abnormal Involuntary Movement Scale (AIMS; total score, Q8 score)

CONTACTS AND LOCATIONS:
Overall Officials: David Coghill, ', Principal Investigator — University of Dundee
Locations (4):
- Zentralinstitut fuer seelische gesundheit, Mannheim, Stadtkreis, Germany
- Vadaskert Child and Adolescent Psychiatry Hospital and Outpatient Clinic, Budapest, Hungary
- Universita degli Studi di Cagliari, Cagliari, Sardinia, Italy
- University of Dundee, Dundee, Tayside, United Kingdom

REFERENCES:
- [Derived] Inglis SK, Carucci S, Garas P, Hage A, Banaschewski T, Buitelaar JK, Dittmann RW, Falissard B, Hollis C, Kovshoff H, Liddle E, McCarthy S, Nagy P, Neubert A, Rosenthal E, Sonuga-Barke E, Wong I, Zuddas A, Coghill DC; ADDUCE Consortium. Prospective observational study protocol to investigate long-term adverse effects of methylphenidate in children and adolescents with ADHD: the Attention Deficit Hyperactivity Disorder Drugs Use Chronic Effects (ADDUCE) study. BMJ Open. 2016 Apr 26;6(4):e010433. doi: 10.1136/bmjopen-2015-010433. PMID 27118284